CLINICAL TRIAL: NCT06717893
Title: Clinical and Laboratory Characteristics of a Population of Children and Adolescents With Newly Diagnosed Type 1 Diabetes and Insulin Requirements at Onset
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: ESORD1T
Record Dates: First submitted 2024-12-01; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-10

CONDITIONS: Type 1 Diabetes (T1D)
Keywords: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The clinical implication of this study lies in the identification of factors that may predict reduced insulin sensitivity in children and adolescents at the onset of Type 1 Diabetes and would help the physician to undertake appropriate therapy more quickly by achieving the correct therapeutic dosage, in order to achieve good metabolic compensation at an early stage and thus reduce the time (and costs) of hospitalisation.

DETAILED DESCRIPTION:
The primary aim of this observational, retrospective, single-centre, non-pharmacological study is to assess whether the presence of clinical and laboratory predictive factors at the onset of type 1 diabetes may be related to an increased insulin requirement in a population of pediatric and adolescent patients with diagnosis of type 1 diabetes between January 2014 and December 2018 at the Pediatrics Unit of the IRCCS Azienda Ospedaliero-Universitaria of Bologna, Italy. The secondary aim is to assess the insulin requirement 1 year after the onset of type 1 diabetes. This study consists of collection and analyses of clinical and laboratory data of patients enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Age ≤ 14 years at the time of diagnosis of type 1 diabetes;
* Diagnosis of type 1 diabetes confirmed between January 2014 and December 2018 at the Pediatrics Unit of the IRCCS Azienda Ospedaliero-Universitaria of Bologna, Italy;
* Patients with at least 1 year of follow-up after diagnosis od type 1 diabetes;
* Obtaining informed consent from parents/legal guardian of pediatric patients.

Exclusion Criteria:

* Patients with diabetes other that type 1;
* Patients followed at other centres at the time of onset of type 1 diabetes.

Max Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric and adolescent patients with type 1 diabetes onset between January 2014 and December 2018, with age ≤ 14 years at the time of diagnosis, and who referred to the Pediatrics Unit of the IRCCS Azienda Ospedaliero-Universitaria of Bologna, Italy.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2020-10-09 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Insulin requirement | at onset of type 1 diabetes, 3 months, and 12 months
  maximum amount of insulin administered subcutaneously during hospitalisation per kg of body weight in 24 hours (U/kg/die)
Laboratory data | at onset of type 1 diabetes, 3 months, and 12 months
  glucose; total cholesterol; HDL cholesterol; triglycerides (mg/dL)

CONTACTS AND LOCATIONS:
Overall Officials: Giulio Maltoni, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy